CLINICAL TRIAL: NCT03873467
Title: Efficacy of an Evidence-based Healthy Lifestyle Intervention for People Following CVA
Brief Title: Group Lifestyle Balance™ for Individuals With Stroke (GLB-CVA)
Acronym: GLB-CVA
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Baylor Research Institute (Other)
Collaborators: National Institute on Disability, Independent Living, and Rehabilitation Research (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: BSWRI 018-714
Record Dates: First submitted 2019-03-07; First posted 2019-03-13 (Actual); Last update posted 2025-10-08 (Actual); Status verified 2025-10

CONDITIONS: Stroke
Keywords: Group Lifestyle Balance; Physical Activity; Stroke; Weight-loss; Dietary Behaviors
MeSH Terms: conditions — Stroke; Motor Activity; Weight Loss

STUDY DESIGN:
Intervention Model Description: Randomized Controlled Trial (RCT). Participants will be randomized into one of two groups: (1) the GLB Intervention Group and (2) the wait-list controlled group.
Who Masked: Outcomes Assessor
Masking Description: Outcomes Assessor will be masked to group allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- GLB Weight-Loss Intervention (Experimental): The GLB program, adapted for individuals with stroke, will be delivered to participants over a 12-month period, divided into 22 in-person or virtual, group sessions. The intervention promotes 5-7% weight-loss by reducing calories and increasing exercise (150 minutes of moderate physical activity per week).
  Interventions: Behavioral: Group Lifestyle Balance
- Wait-List Control (Other): The wait-list control group will receive no intervention for 6 months after enrollment. After the 6 month control period, the wait-list control group will receive the GLB Intervention.
  Interventions: Other: Usual Care

INTERVENTIONS:
Behavioral: Group Lifestyle Balance — The Group Lifestyle Balance (GLB) program is a self-management intervention that has been shown to result in weight-loss and reduce the risk for Type 2 diabetes through increased physical activity and healthy eating behaviors in the general population. The GLB is a direct adaptation of the Diabetes Prevention Program, both developed at the Diabetes Prevention and Support Center at the University of Pittsburgh. The GLB is designed for delivery in a group-based, community setting, and has resulted in weight-loss in a variety of settings, such as community centers, churches, worksites, and healthcare systems. The GLB curriculum used in this study has been adapted for people with stroke.
  Arms: GLB Weight-Loss Intervention
Other: Usual Care — Participants randomized to the wait-list control group will receive usual care for 6 months before beginning the modified GLB program.
  Arms: Wait-List Control

SUMMARY:
The purpose of this RCT is to examine the efficacy of the Group Lifestyle Balance (GLB) program adapted for people with stroke (CVA) on primary (weight) and secondary outcomes at 3, 6, 12 months from enrollment into the program.

DETAILED DESCRIPTION:
Weight gain greatly increases the risk of chronic diseases after stroke such as diabetes, metabolic syndrome, pulmonary and heart disease. Approaches to weight-loss are lacking, yet necessary, due to the unique physiological and cognitive needs of persons with CVA. There is evidence that interventions that improve physical activity and healthy eating behaviors concurrently offer greatest potential for weight-loss. The Group Lifestyle Balance (GLB) intervention is a 12-month, evidence-based weight-loss program that has been used extensively with the general population, but not with people after CVA. Investigators modified the program to meet the needs of people post stroke (GLB-CVA).

Study Aims:

The study consists of five specific aims.

Specific Aim 1: To create an appropriate adaptation of the DPP-GLB program that meets the unique needs of people post CVA (GLB-CVA) using a Community-Based Participatory Research approach and Advisory Board of key stakeholders (patients, caregivers, clinicians, researchers).

Specific Aim 2: To establish the feasibility of delivering the GLB-CVA intervention.

Specific Aim 3: Conduct a randomized controlled trial (RCT) to examine the effectiveness of the GLB-CVA on primary and secondary outcomes in the intervention group compared to the wait-list control group at 3, 6, and 12 months from baseline.

Specific Aim 4: Describe the effect of the GLB-CVA on metabolic biomarkers in the experimental group compared to the wait-list control group at baseline, 3, and 6 months.

Specific Aim 5: Describe the association between biomarkers of neurodegeneration and physiologic, functional, and patient reported outcomes at baseline, 3, and 6 months.

ELIGIBILITY:
Inclusion Criteria:

* 18 to 85 years of age
* BMI ≥25
* All types of stroke
* At least 12 months post first stroke
* Physician approval

Exclusion Criteria:

* Low cognition
* Not fluent in the English language
* Conditions for which physical activity is contraindicated
* Taking medication for type 2 diabetes
* Residing in a hospital, acute rehabilitation setting, or skilled nursing facility
* Pregnancy
* Pre-existing diagnosis of an eating disorder

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2019-07-08 (Actual); Primary Completion 2022-12-30 (Actual); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Change in weight | Baseline, 3, 6, 12 months
  Will be obtained using the same scale over the study period that is accessible to people with and without a mobility device (e.g., walker; wheelchair).

SECONDARY OUTCOMES:
Physical Activity | Baseline, 3, 6, 12 months
  Accelerometers will be worn by participants for two weeks around each study visit to objectively track physical activity participation (amount and intensity). Participants will be given the Actigraph accelerometer at the beginning of the study and will be provided with verbal and written instructions.
Arm Circumference | Baseline, 3, 6, 12 months
  Arm circumference measured at mid-upper arm following ACSM guidelines. A total of three measurements will be taken and an average of the three will be used. Measurements will be taken in centimeters.
Blood Pressure | Baseline, 3, 6, 12 months
  Using an automatic cuff (average of three readings, patient seated) diastolic and systolic scores will be recorded
Cholesterol | Baseline, 3, 6, 12 months
  Fasting venous sample will be obtained. Coordinators are trained phlebotomists.
Risk of Diabetes | Baseline, 3, 6, 12 months
  The Framingham Heart Study diabetes risk score will be calculated using predictors including age, gender, fasting glucose, BMI, HDL cholesterol and triglyceride levels, blood pressure, and parental history. Risk score calculator and regression model are free and used in GLB weight-loss trials. Risk score calculator and regression model are free and used in GLB weight-loss studies. Each risk predictor is assigned points ranging from 2-10. Risk factors are combined and a total score is calculated, with higher scores designating greater 8-year risk.The age range for this score is 45 years to 64 years, and therefore only individuals within this age will have calculated scores. Furthermore, the minimum cut-off score is 3.
10 Meter Walk Test (10MWT) | Baseline, 3, 6, 12 months
  Assesses walking speed in (m/s) which is correlated to mobility in the community, capacity to perform ADLs, risk of falls, re-hospitalization, and risk of cognitive decline.
6 Minute Walk Test (6MWT) | Baseline, 3, 6, 12 months
  Assesses distance walked over 6 minutes as a sub-maximal test of aerobic capacity. Endurance is essential to participate in community-based activities.
Perceived Social Support | Baseline and 12 months
  The Multidimensional Scale of Perceived Social Support (MSPSS) is comprised of 12 questions with a 4-item subscale. The MSPSS is designed to assess perception of social support from friends, family, and significant others
Self-reported activities of health using the Self-Rated Abilities for Health Practice scale | Baseline and 12 months
  Measure includes 28 items that assess health practices among people with disabilities and yields a total Health Practices score plus 4 subscales scores regarding Exercise, Nutrition, Health Practices, and Psychological Well Being. Items are rated on a 5-point scale from 0 'not at all' to 4 'completely.' Scores range from 0-28 with higher scores indicating higher exercise self-efficacy.
Neighborhood walkability using Walk Score® | Baseline
  Walk Score® is publicly available and measures the walkability of any address using a patented system. For each address, Walk Score ® analyzes hundreds of walking routes to nearby amenities and awards points based on distance to each amenity. Walk Score® also measures pedestrian friendliness by analyzing population density and road metrics such a block length and intersection density. Scores are given on a scale of 0 to 100.
Resting Metabolic Rate | Baseline
  MedGem® is an FDA cleared and validated indirect calorimetry device. It is handheld and measures oxygen consumption (V02) to determine resting metabolic rate (RMR).
Behavioral Risk Factor Surveillance | Baseline, 3, 6, 12 months
  The BRFSS is a state-based system of health surveys that collects information on health risk behaviors, preventative health practices, and health care access primarily related to chronic disease and injury. The GLB-TBI uses the two subscales of Healthy Eating and Physical Activity from the 2017 version of the BRFSS. It consists of 14 items.
Participant quality of ife | Baseline, 6, 12 months
  Quality of life will be assess using the stroke impact scale (SIS), which assesses 8 dimensions of health-related QOL specific to people post CVA including subscales (using a 5pt Likert scale) assessing strength, memory and thinking, emotion, communication, activities of daily living, mobility, hand function, and participation/role function
Stressful Life Events using the Holmes and Rahe Stress Inventory | Baseline and 12 months
  This inventory consists of 40 life events and asks the participant to recall if any of the events happened within the previous year (e.g., death of spouse; personal illness; change in sleep). Endorsement of these events are totaled and higher scores indicate a greater amount of stressful life events. Point values for the Holmes and Rahe Stress Inventory were weighted and summed for each individual based on scoring instructions. Individuals who scored 150 points or less were categorized as low susceptibility to a health breakdown in the next two years, 151-300 points were 50% chance of health breakdown, and 301 points or more were 80% chance of health breakdown.
Executive Function and Cognition using the Montreal Cognitive Assessment | Baseline, 3, and 12 months
  The MOCA is a brief, 8-section assessment of various cognitive domains including executive function, memory, language, attention, concentration, orientation, and working memory in neurologic populations.Each item on the MOCA is allocated a set of points adding up to 30.
Habit Formation | Baseline, 3, and 12 months
  The self-reported habit index (SRHI) measures the self-reported perceptions of habit strength for an identified behavior. It consists of 12 items for each selected behavior and uses a 7-point Likert scale from "completely disagree" to "completely agree." Higher totals represent greater perception of habit strength. The SRHI showed high reliability across four studies with alphas of .89, .92, .89, .94, .95, .94, and .85.
Stroke Severity | Baseline
  The Modified Rankin Scale (MRS) measures the degree of disability or dependence for daily activities of people who have had a stroke. The MRS is an ordinal scale with six categories ranging from zero (no symptoms) to five (complete physical dependence). A score of six signifies death.
Pain Interference | Baseline, 3, 6, and 12 months
  The Pain Interference-Short Form is taken from the Patient-Reported Outcomes Measurement Information System (PROMIS). This measure is used to assess adult self-reported consequences of pain and pain consequences (e.g. interference in social, cognitive, emotional, physical and recreational activities). This measure consists of four questions with five response option ranging from one to five. The sum of all responses creates a total raw score. This measure is normed to the US general population.
Sleep Disturbance | Baseline, 3, 6, 12 months
  The Sleep Disturbance-Short Form 4a is taken from the Patient-Reported Outcomes Measurement Information System (PROMIS) and used to assess adult sleep disturbance profiles. This measure has four questions, each with five response options ranging in value from one to five. The sum of each response creates a total raw score. The measure is normed to the US general population.
Waist Circumference | Baseline, 3, 6, and 12 months
  Waist circumference will be measured at the umbilicus following ACSM guidelines. A total of three measurements will be taken and an average of the three will be the final measurement used. Measurements will be scored in centimeters.
HbA1c | Baseline, 3, 6, and 12 months
  Fasting venous sample will be obtained for hemoglobin a1c to assess average blood sugar level over the past 2-3 months. Coordinators are trained phlebotomists.
Triglycerides | Baseline, 3, 6, 12 months
  Fasting venous sample will be obtained. Coordinators are trained phlebotomists.
Blood Glucose | Baseline, 3, 6, 12 months
  Fasting venous sample will be obtained. Coordinators are trained phlebotomists.
Biomarker Analysis | Baseline, 3, and 6 months
  Isrin, Angiogenic factors (VEGF), Total Homocysteine, Lipoprotein-associated phospholipase A2 (Lp-PLA2), ICF-1, Brain derived neurotrophic factor (BDNF), and Tau proteins (total and phosphorylated) will be drawn to assess relationships with outcome variables.
Stages of Change | Baseline, 3, 6, and 12 months
  A modified version of Prochaska and DiClemente's Stages of Change model will be administered to measure readiness for behavior change. The measure consists of two behaviors (eating and exercise) with five questions each related to a stage of change (precontemplation, contemplation, preparation, action, maintenance).
Metabolic Score Calculator (MetS) | Baseline, 3, 6, and 12 months
  The metabolic score calculator will be used at all time points to determine the risk for metabolic syndrome. The following variables will be used to determine metabolic risk using the free metabolic risk calculator: gender, race and ethnicity, systolic blood pressure, fasting glucose, triglycerides, high-density lipoprotein (HDL), weight, height, and waist circumference. Scores are calculated are standardized to the general population.
CRISIS (CoRonavIruS Health Impact Survey) V0.3 Adult Baseline Form | Up to 12 months
  This self-report survey was developed by the National Institute of Mental Health. The full survey consists of 64 questions with an open-ended section at the end to elicit concerns and feedback related to the effects of COVID-19. For this current study, however, only sections on Exposure Status (10 items), Life Changes (15 items), and Emotions/Worries (7 items), and the open-ended question will be asked. Questions are asked "over the past two weeks."
PROMIS Social Isolation Short Form 4a | Up to 12 months
  The Social Isolation Short-Form 4a is taken from the Patient-Reported Outcomes Measurement Information System (PROMIS). This form assesses the perceptions of being "avoided, excluded, detached, disconnected from, or unknown by, others. There is no timeframe for the form. The measure is normed to the US population.
Media Questionnaire | Up to 12 months
  To assess media exposure and fear of media exposure during COVID-19 we have added 6 questions. These are asked "over the past two weeks." These questions address time spent watching the television, listening to radio, reading the newspaper, and searching the internet and social media. In addition, a 6th question related to fear is asked using a 5-point Likert scale.

CONTACTS AND LOCATIONS:
Overall Officials: Simon J Driver, PhD, Principal Investigator — Baylor Scott & White Institute for Rehabilitation (BSWIR)
Locations (1):
- Baylor Scott & White Institute for Rehabilitation, Dallas, Texas, United States

REFERENCES:
- [Background] Driver S, McShan E, Swank C, Grobe K, Calhoun S, Bailey R, Kramer K. Creating an appropriate adaptation of a healthy lifestyle intervention for people after stroke. Brain Inj. 2020 Sep 18;34(11):1497-1503. doi: 10.1080/02699052.2020.1808703. Epub 2020 Aug 19. PMID 32813569
- [Background] Driver S, Swank C, Froehlich-Grobe K, McShan E, Calhoun S, Bennett M. Weight Loss After Stroke Through an Intensive Lifestyle Intervention (Group Lifestyle Balance-Cerebrovascular Accident): Protocol for a Randomized Controlled Trial. JMIR Res Protoc. 2019 Oct 18;8(10):e14338. doi: 10.2196/14338. PMID 31628790